CLINICAL TRIAL: NCT04354779
Title: Antikörperseroprävalenz Und Hintergrundinfektionsrate Von SARS-CoV-2 in Einem österreichischen Schlüsselkollektiv an Arbeitnehmer*Innen
Brief Title: Antibody Seroprevalence and Rate of Asymptomatic Infections With SARS-CoV-2 in Austrian Hospital Personnel.
Status: Completed | Type: Observational
Sponsor: AUVA (Other)
Collaborators: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Wolfgang Schaden, Principal Investigator, AUVA
Other Study IDs: AUVA SARS-CoV-2 Studie
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2; SARS-CoV 2; Coronavirus Infection; Covid19
Keywords: COVID-19 diagnostic testing; SARS-CoV 2; Severe Acute Respiratory Syndrome Coronavirus 2
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AUVA HCW: health care workers in Austrian trauma hospitals and rehabilitation facilities of the Austrian Social Insurance for Occupational Risks (AUVA)
  Interventions: Diagnostic Test: a specifically designed self-administered questionnaire

INTERVENTIONS:
Diagnostic Test: a specifically designed self-administered questionnaire — The questionnaire consists of the following items: questions related to personal health, traveling activities, living situation, as well as inquiries of symptoms and comorbidities.

SUMMARY:
Context: On March 11, the World Health Organization (WHO) announced the current corona virus disease 2019 (COVID-19) outbreak as a pandemic. The first laboratory-confirmed case of COVID-19 in Austria was announced on February 27, 2020. Since then, the incidence of infection follows a gradual increase. Measurements taken by the Austrian government include travel restrictions, closing of national borders, social distancing, a mandatory use of facemasks in public, and closing of stores and restaurants. The underlying aim of those imposed restrictions is to contain the viral transmission and to slow spreading of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

Objectives: The aims of this study are to determine i) how many employees in Austrian trauma hospitals and rehabilitation facilities have virus specific IgG and IgM antibodies against SARS-CoV-2, ii) how many are active virus carriers (symptomatic and asymptomatic), iii) how many employees are in their incubation period during the study period, and iv) to calculate the SARS-CoV-2 prevalence together with a specific occupation associated infection risk within the different specifications of health care workers.

Study Design: Open uncontrolled observational cross-sectional study.

Setting/Participants: A total of 4000 employees in 11 Austrian trauma hospitals and rehabilitation facilities of the Austrian Social Insurance for Occupational Risks (AUVA) will be invited to participate in the study.

Study Interventions and Measures: An antibody test for SARS-CoV-2 specific IgG and IgM antibodies, and a RT-PCR test based on oropharyngeal swab samples, as well as laboratory-based antibody tests using ELISA, will be implemented to ensure protection and preservation of health in hospital staff and are not part of the study. The tests will be conducted twice, with approximately two weeks in between testing. The results of the tests will be used for statistical analysis in this study together with a questionnaire including questions related to personal health, traveling activities, living situation, as well as inquiries of symptoms and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* employees in Austrian trauma hospitals and rehabilitation facilities of the Austrian Social Insurance for Occupational Risks (AUVA)

Exclusion Criteria:

* NA

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All employees in Austrian trauma hospitals and rehabilitation facilities of the Austrian Social Insurance for Occupational Risks (AUVA) will be invited to participate in the study. In total, 4000 individuals in 12 hospitals and rehabilitation facilities in Austria will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 3301 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-08-23 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Antibody status in HCW | 4 months
  To determine how many employees in Austrian trauma hospitals and rehabilitation facilities have already virus specific IgG and IgM antibodies against SARS-CoV-2.
Active virus carriers in HCW | 4 months
  To determine how many are actively infected with or without showing symptoms.
Incubation time | 4 months
  To determine how many employees are in their incubation period during study time.

SECONDARY OUTCOMES:
Background incidence rate | 4 months
  To evaluate the "background incidence rate" of COVID-19 to calculate the SARS-CoV-2 prevalence in a defined cohort of the Austrian population.
Occupation associated infection risk | 4 months
  To calculate a specific occupation associated infection risk within the different specifications of health care workers amongst AUVA employees.

CONTACTS AND LOCATIONS:
Locations (1):
- Allgemeine Unfallversicherungsanstalt, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
IPD will be encrypted and anonymised.